CLINICAL TRIAL: NCT02298335
Title: A Prospective Observational Study to Assess the Efficacy an Safety of Glucocorticoid Therapy in the Treatment of Adult Idiopathic Nephrotic Syndrome
Brief Title: Glucocorticoid in Treatment of Adult Idiopathic Nephrotic Syndrome：a Prospective Observational Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, MD, Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1401
Record Dates: First submitted 2014-10-20; First posted 2014-11-21 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Nephrotic Syndrome，Idiopathic
Keywords: Prednisone; idiopathic nephrotic syndrome; prospective
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- prednisone (Experimental): First,full-dose induction period, then protracted tapering period.
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: prednisone — Full-dose induction period: Prednisone 1mg/kg.day, maximum 60mg/day, orally, divided into 3 times; Protracted tapering period: orally, no ask for fract. dos.

SUMMARY:
This study is to assess the efficacy and safety of 8-weeks full-dose induction protocol (prednisone 1mg/kg, maximum 60mg/day) and protracted tapering protocol in the treatment of adult idiopathic nephrotic syndrome.

DETAILED DESCRIPTION:
In full-dose induction period, patients scheme to visit at the 4th and 8th week, and in protracted tapering period at 10th , 22nd, 42nd and 66th week. If the patients reach complete remission within 4 weeks, prednisone may be decreased at the 6th week, otherwise keep on the course to the 8th week. All patients reach complete remission will shift to protracted tapering period and follow up until prednisone withdrawal, except the cases that relapse and drop out the study. If proteinuria reappears in someone, angiotensin-converting enzyme inhibitor（ACEI） or angiotensin receptor blocker（ARB） will be considered combination, on the premise of the blood pressure is affordable.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed written informed consent form
* Age between 18-65 years, female or male
* Patients with diagnosis of nephrotic syndrome ( proteinuria ≥3.5 g/24h, and serum albumin ≤30g/L ),
* Pathological diagnosis with minimal change disease (MCD), focal segmental glomerulosclerosis (FSGS) and podocyte disease
* Serum creatinine < 3mg/dl ( 265.2umol/L), estimated glomerular filtration rate(eGFR) no less than 30 ml/min.1.73 m2

Exclusion Criteria:

* Patients who didn't sign written informed consent form
* Patients who have received full-dose prednisone treatment for more than 2 weeks, or pulsed methylprednisolone (>7.5mg/kg.day) within 2 weeks
* Patients who have taken immunosuppressants within 3 months, as Cyclosporine A, Tacrolimus, Mycophenolate Mofetil, Cyclophosphamide, or Leflunomide etc.
* Patients who have impaired liver function, with Alanine aminotransferase(ALT) or Aspartate aminotransferase(AST) twice more than the normal upper limit, or who have viral hepatitis B with hepatitis B e antigen(HBeAg) positive or hepatitis B virus DNA (HBV-DNA) reduplicative
* Patients who have contraindications to glucocorticoid, for example diabetes, obesity (BMI>28kg/m2 before disease onset), femoral head necrosis, or active infection.
* Patients who have family history of kidney disease
* Patients who have definite secondary facts of this disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2014-05-13; Primary Completion 2019-07 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
the cumulative complete remission rate of 8-weeks full-dose induction protocol | 8 weeks

SECONDARY OUTCOMES:
the relapse rate of complete remission participants protracted tapering protocol | 66 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD, Study Chair — Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Nanjing, Jiangsu, China